CLINICAL TRIAL: NCT04337827
Title: Phase II Study of Rituximab and Acalabrutinib in Newly Diagnosed B Cell Post Transplant Lymphoproliferative Disorder (PTLD)
Brief Title: Rituximab and Acalabrutinib in Newly Diagnosed B Cell Post Transplant Lymphoproliferative Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Deepa Jagadeesh (Other)
Responsible Party: Sponsor-Investigator, Deepa Jagadeesh, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3419
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Post-transplant Lymphoproliferative Disorder
MeSH Terms: interventions — Rituximab; acalabrutinib; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rituximab and Acalabrutinib (Experimental): Participants will receive treatment of Rituximab weekly for 4 weeks, and Acalabrutinib twice daily for 4 weeks. Response assessment via diagnostic CT scans will dictate further treatment decisions.
  Interventions: Drug: Rituximab; Drug: Acalabrutinib; Diagnostic Test: CT scans

INTERVENTIONS:
Drug: Rituximab — Weekly x 4 weeks.
  If diagnostic test reveals complete response, then participant will continue with one additional 28 day cycle. If partial response, then proceed with 3 additional 28 day cycles. If stable disease or progression of disease, then go off study treatment and proceed onto Long Term Follow Up (LTFU).
  Other Names: Rituxan; Mabthera
Drug: Acalabrutinib — 100mg twice per day (BID) x 4 weeks (28 day cycle)
  If diagnostic test reveals complete response, then participant will continue with one additional 28 day cycle. If partial response, then proceed with 3 additional 28 day cycles. If stable disease or progression of disease, then go off study treatment and proceed onto LTFU.
  Other Names: ACP-196
Diagnostic Test: CT scans — 2 weeks (day 36 ± 5 days) after end of cycle 1 treatment.

SUMMARY:
The purpose of this study is to evaluate how effective rituximab and acalabrutinib are when given as a combination treatment for newly diagnosed B cell post transplant lymphoproliferative disorder (PTLD). Currently there is no approved therapy for PTLD. Rituximab alone is commonly used and works in some cases, but not others. In addition, participants with PTLD have trouble tolerating therapies with large amounts of side effects due to their health conditions and medications for their transplant. Due to these reasons the study team is looking for a new treatment with novel targeted agents in order to improve outcomes and to minimize toxicity.

Based on emerging data of clinical efficacy of acalabrutinib in B cell malignancies and an unmet need for novel therapies in PTLD, this study will investigate the use of rituximab and acalabrutinib in participants with newly diagnosed B cell PTLD.

DETAILED DESCRIPTION:
This is a non-randomized phase II study of acalabrutinib plus rituximab in newly diagnosed B-cell PTLD in participants with both solid organ transplant (SOT) and Bone marrow transplant (BMT).

Acalabrutinib is an inhibitor of Bruton Tyrosine Kinase (BTK). BTK is important in B cells and plays a role in the development of PTLD. Acalabrutinib is approved in the US for the treatment of adult participants with indolent lymphoma, mantle cell lymphoma, and is being evaluated to treat other lymphomas.

Rituximab has been approved for treatment of B cell non-Hodgkin lymphoma (NHL). While not approved for PTLD, it has become the mainstay of treatment.

The primary objective of this study is to determine the overall response rate to combination treatment with rituximab and acalabrutinib in patients with PTLD.

The secondary objectives of this study is to determine response rates, survival, failure rates, and safety elements in participants with PTLD treated with combination rituximab and acalabrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a biopsy confirmed newly diagnosed CD20 positive B cell PTLD.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. ECOG 3 will be permitted if the decline in performance status is due to lymphoma. [See Appendix 1]
* Subjects must have adequate hematologic, hepatic, and renal function as defined below:

  * Hemoglobin ≥ 8 gm/dL
  * Absolute neutrophil count ≥500/mcL (unless documented bone marrow involvement with lymphoma)
  * Platelet count ≥50000/mcL (unless there is documented bone marrow involvement with lymphoma)
  * Prothrombin time/international normalized ratio (INR) or activated partial thromboplastin time (aPTT) (in the absence of Lupus anticoagulant) < 2x ULN.
  * Total bilirubin ≤1.5X upper limit of normal (ULN)
  * Creatinine ≤2.5X upper limit of normal (ULN)
  * Alanine aminotransferase/aspartate aminotransferase (ALT/AST) < 2.5 X or ≤5X ULN for patients with document hepatic involvement with lymphoma
* Women of childbearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) during treatment and for 12 months after last dose of study treatment. Women who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential.
* Subjects must be willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
* Subjects must have the ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria:

* Prior treatment with any BTK inhibitor
* Subjects receiving any other investigational agents or participating in another therapeutic clinical trial.
* Subjects with active (treated or untreated) brain metastases/ central nervous system (CNS) disease (including but not limited to CNS PTLD) will be excluded from this clinical trial
* Prior malignancy (or any other malignancy that requires active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, early stage prostate cancer or other cancer from which the subject has been disease free for ≥ 3 years
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll in the study.
* Has difficulty with or is unable to swallow oral medication, or has significant gastrointestinal disease that would limit absorption of oral medication.
* Known history of infection with HIV. HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with acalabrutinib.
* Patients with uncontrolled concurrent illness like active infection (eg, bacterial, viral, or fungal) requiring IV antibiotics or psychiatric illness/social situations that would limit compliance with study requirements
* Known history of drug-specific hypersensitivity or anaphylaxis to acalabrutinib or rituximab (including active product or excipient components).
* Active bleeding, history of bleeding diathesis (eg, hemophilia or von Willebrand disease).
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon)
* Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
* History of significant cerebrovascular disease or event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug.
* Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
* Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded.
* History of progressive multifocal leukoencephalopathy (PML)
* Breastfeeding or pregnant. Pregnant or breastfeeding women are excluded from this study because it is unknown how acalabrutinib and rituximab can affect the fetus or infant. Rituximab can cross the placenta and is found in breast milk. Acalabrutinib has been found in the breast milk of animals and there is not significant data regarding its effect during pregnancy.
* Vaccination with live virus vaccines is not allowed within 4 weeks of study treatment of or during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Jagadeesh, MD, MPH, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual patient data in order to protect the confidentiality of the subjects who enroll on this study

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab and Acalabrutinib: Participants will receive treatment of Rituximab weekly for 4 weeks, and Acalabrutinib twice daily for 4 weeks. Response assessment via diagnostic CT scans will dictate further treatment decisions.
  Rituximab: Weekly x 4 weeks.
  If diagnostic test reveals complete response, then participant will continue with one additional 28 day cycle. If partial response, then proceed with 3 additional 28 day cycles. If stable disease or progression of disease, then go off study treatment and proceed onto Long Term Follow Up (LTFU).
  Acalabrutinib: 100mg twice per day (BID) x 4 weeks (28 day cycle)
  If diagnostic test reveals complete response, then participant will continue with one additional 28 day cycle. If partial response, then proceed with 3 additional 28 day cycles. If stable disease or progression of disease, then go off study treatment and proceed onto LTFU.
  CT scans: 2 weeks (day 36 ± 5 days) after end of cycle 1 treatment.
Period: Overall Study
Arm/Group | Rituximab and Acalabrutinib
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR will be estimated along with 90% Confidence Intervals (CIs), and compared against the null using exact binomial test. Logistic regression model will be used to identify factors associated with response status.
Time Frame: Up to 8 weeks after treatment
Population: Sponsor terminated financial support of all research activity not associated with active subjects receiving study medication enrolled under this IND, it has been decided to close enrollment and to cease long-term follow-up of subjects. Zero participants were followed past the end of treatment for several reasons, including removal of funding that prevented follow-up or participants reaching stable disease (per protocol, participant does not get followed). Therefore, no data was collected.
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as all patients that achieve a CR based on end of treatment scans, using the Lugano Criteria
Time Frame: at 6 months after treatment
Population: Due to notification by AstraZeneca to terminate financial support of all research activity not associated with active subjects receiving study medication enrolled under this IND, it has been decided to close the study to enrollment and to cease long-term follow-up of subjects not actively receiving study medication. Participants were unable to be followed after the end of treatment for 6 months; therefore, no data was collected.
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as all patients that achieve a CR based on end of treatment scans, using the Lugano Criteria
Time Frame: at 12 months after treatment
Population: Due to notification by AstraZeneca to terminate financial support of all research activity not associated with active subjects receiving study medication enrolled under this IND, it has been decided to close the study to enrollment and to cease long-term follow-up of subjects not actively receiving study medication. Participants were unable to be followed after the end of treatment for 12 months, therefore, no data was collected.
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as all patients that achieve a CR based on end of treatment scans, using the Lugano Criteria
Time Frame: at 24 months after treatment
Population: Due to notification by AstraZeneca to terminate financial support of all research activity not associated with active subjects receiving study medication enrolled under this IND, it has been decided to close the study to enrollment and to cease long-term follow-up of subjects not actively receiving study medication. Participants were unable to be followed after the end of treatment for 24 months, therefore, no data was collected.
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Partial Response Rate (PRR)
Description: PRR is defined as all patients that achieve a PR based on end of treatment scans, using the Lugano Criteria.
Time Frame: at 6 months after treatment
Population: as for outcome 2
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Partial Response Rate (PRR)
Description: PRR is defined as all patients that achieve a PR based on end of treatment scans, using the Lugano Criteria.
Time Frame: at 12 months after treatment
Population: as for outcome 3
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Partial Response Rate (PRR)
Description: PRR is defined as all patients that achieve a PR based on end of treatment scans, using the Lugano Criteria.
Time Frame: at 24 months after treatment
Population: Due to notification by AstraZeneca to terminate financial support of all research activity not associated with active subjects receiving study medication enrolled under this IND, it has been decided to close the study to enrollment and to cease long-term follow-up of subjects not actively receiving study medication. Participants were unable to be followed after the end of treatment for 24 months; therefore, no data was collected.
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

8. Secondary Outcome: Duration of Response (DOR)
Description: DOR is only measured in responders. DOR is defined as the time from documented response (CR or PR) to the time of confirmed disease progression or death due to any cause, whichever occurs first. Subjects who are still alive and free from progression at the time of data cutoff date, lost to follow-up, have discontinued study, or have initiated other non-protocol anti-tumor therapy (NPT) will be censored at the last tumor assessment when subjects are progression-free.
Time Frame: Up to 3 years after treatment
Population: Due to notification by AstraZeneca to terminate financial support of all research activity not associated with active subjects receiving study medication enrolled under this IND, it has been decided to close the study to enrollment and to cease long-term follow-up of subjects not actively receiving study medication. Participants were unable to be followed after the end of treatment for 3 years; therefore, no data was collected.
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

9. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS as defined as the time from first dose to documented disease progression, or death from any cause, whichever occurs first. Data for subjects who are still alive and free from progression at the time of data cutoff date, lost to follow-up, have discontinued the study, or have initiated NPT will be censored on last assessment (or, if no post-baseline tumor assessment, at the time of first dose plus 1 day)
  Estimated using Kaplan-Meier method and compared using log-rank test. Cox proportional hazard model will be used to identify factors associated with survival endpoint.
Time Frame: at 6 months after treatment
Population: Due to notification by AstraZeneca to terminate financial support of all research activity not associated with active subjects receiving study medication enrolled under this IND, it has been decided to close the study to enrollment and to cease long-term follow-up of subjects not actively receiving study medication. Participants were unable to be followed after the end of treatment for 6 months, therefore, no data was collected.
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

10. Secondary Outcome: Progression Free Survival (PFS)
Description: as for outcome 9
Time Frame: at 12 months after treatment
Population: Due to notification by AstraZeneca to terminate financial support of all research activity not associated with active subjects receiving study medication enrolled under this IND, it has been decided to close the study to enrollment and to cease long-term follow-up of subjects not actively receiving study medication. Participants were unable to be followed after the end of treatment for 12 months; therefore, no data was collected.
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

11. Secondary Outcome: Progression Free Survival (PFS)
Description: as for outcome 9
Time Frame: at 24 months after treatment
Population: as for outcome 7
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

12. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from first dose to death from any cause. Data for subjects who are still alive at the time of data cutoff date, lost to follow-up, have discontinued the study (or, if no post-baseline assessment, at the time of first dose plus 1 day) will be censored on last assessment
  Estimated using Kaplan-Meier method and compared using log-rank test. Cox proportional hazard model will be used to identify factors associated with survival endpoint.
Time Frame: Up to 3 years after treatment
Population: as for outcome 8
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

13. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is measured from the time from study entry to any treatment failure including discontinuation of treatment for any reason, such as disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death.
Time Frame: Up to 3 years after treatment
Population: as for outcome 8
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With a Grade 3 Adverse Event (AE) or Higher
Description: Safety as defined by number of participants with a grade 3 AE or higher
Time Frame: Up to 3 years after treatment
Population: as for outcome 8
Arm/Group | Rituximab and Acalabrutinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed on all subjects from the point of Eligibility Screening (baseline) to 30 days following the last dose of the study drug (which was 10 months on average).
Arm/Group | Rituximab and Acalabrutinib
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab and Acalabrutinib (N=6)
Lung infection (Infections and infestations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab and Acalabrutinib (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1) — Infections and infestations - Other, specify - COVID
Lung infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Urinary Urgency (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects, unable to perform analysis of data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT04337827/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT04337827/ICF_000.pdf